CLINICAL TRIAL: NCT04091126
Title: A Phase 1, Randomized, Dose and Schedule Evaluation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of Belantamab Mafodotin Administered in Combination With Standard of Care in Participants With Newly Diagnosed Multiple Myeloma
Brief Title: Study of Belantamab Mafodotin Plus Standard of Care (SoC) in Newly Diagnosed Multiple Myeloma
Acronym: DREAMM 9
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 209664; 2023-507060-39 (Registry Identifier: CTIS)
Expanded Access: NCT03763370 (Available)
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: Bortezomib; Lenalidomide; dexamethasone; VRd; Belantamab mafodotin; Newly diagnosed multiple myeloma; RP3D; DREAMM 9
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; Bortezomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: The study will evaluate different doses/dose schedules of belantamab mafodotin in combination with Velcade (bortezomib), Revlimid (lenalidomide), dexamethasone, (VRd) in up to 8 cohorts and will determine the Recommended Phase 3 dose (RP3D).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Cohort 1: belantamab mafodotin 1.9 mg/kg Q3/4W + VRd/Rd (Experimental): Participants will receive 1.9 milligram /kilogram (mg/kg) Q3W dose of belantamab mafodotin on Day 1 of every cycle for the first 8 cycles in combination with VRd and Q4W dose in combination with Rd from cycle 9 onwards.
  Interventions: Drug: Belantamab mafodotin; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone
- Cohort 2: belantamab mafodotin 1.4 mg/kg Q6/8W + VRd/Rd (Experimental): Participants will receive 1.4 mg/kg Q6W dose of belantamab mafodotin on Day 1 of every other cycle for the first 8 cycles in combination with VRd and Q8W dose in combination with Rd from cycle 9 onwards.
  Interventions: Drug: Belantamab mafodotin; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone
- Cohort 3: belantamab mafodotin 1.9 mg/kg Q6/8W + VRd/Rd (Experimental): Participants will receive 1.9 mg/kg Q6W dose of belantamab mafodotin on Day 1 of every other cycle for the first 8 cycles in combination with VRd and Q8W dose in combination with Rd from cycle 9 onwards.
  Interventions: Drug: Belantamab mafodotin; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone
- Cohort 4: belantamab mafodotin 1.0 mg/kg Q3/4W + VRd/Rd (Experimental): Participants will receive 1.0 mg/kg Q3W dose of belantamab mafodotin on Day 1 of every cycle for the first 8 cycles in combination with VRd and Q4W dose in combination with Rd from cycle 9 onwards.
  Interventions: Drug: Belantamab mafodotin; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone
- Cohort 5: belantamab mafodotin 1.4 mg/kg Q3/4W + VRd/Rd (Experimental): Participants will receive 1.4 mg/kg Q3W dose of belantamab mafodotin on Day 1 of every cycle for the first 8 cycles in combination with VRd and Q4W dose in combination with Rd from cycle 9 onwards.
  Interventions: Drug: Belantamab mafodotin; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone
- Cohort 6: belantamab mafodotin 1.4mg/kg cycle 1, 1.0 mg/kg Q9/12W Cycle 4+VRd/Rd (Experimental): Based on emerging data from Cohort 2-5, participants will receive 1.4 mg/kg dose of belantamab mafodotin on Day 1 of cycle 1, followed by 1.0 mg/kg dose on Day 1 of every third cycle from cycle 4 onwards, in combination with VRd for the first 8 cycles and in combination with Rd from cycle 9 onwards.
  Interventions: Drug: Belantamab mafodotin; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone
- Cohort 7: belantamab mafodotin 1.9 mg/kg Cycle 1, 1.4 mg/kg Q9/12W Cycle 4+VRd/Rd (Experimental): Based on emerging data from Cohort 2-5, participants will receive 1.9 mg/kg dose of belantamab mafodotin of cycle 1, followed by 1.4 mg/kg on Day 1 of every third cycle from cycle 4 in combination with VRd for the first 8 cycles and in combination with Rd from cycle 9 onwards.
  Interventions: Drug: Belantamab mafodotin; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone
- Cohort 8a : belantamab mafodotin 1.9 mg/kg Cycle 1,4; 1.4 mg/kg Q9/12W from Cycle 7 +VRd/Rd (Experimental): Based on emerging data from Cohort 6-7, participants will receive 1.9 mg/kg dose of belantamab mafodotin on Day 1 of cycle 1 and cycle 4, followed by 1.4 mg/kg on Day 1 of every third cycle from cycle 7 onwards, in combination with VRd for the first 8 cycles and in combination with Rd from cycle 9 onwards.
  Interventions: Drug: Belantamab mafodotin; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone
- Cohort 8b: belantamab mafodotin 1.4 mg/kg Cycle 1,3; 1.0 mg/kg Q9/12W from Cycle 6 +VRd/Rd (Experimental): Based on emerging data from Cohort 6-7, participants will receive 1.4 mg/kg IV dose of belantamab mafodotin on Day 1 of cycle 1 and cycle 3, then 1.0 mg/kg on Day 1 of every third cycle from cycle 6 in combination with VRd for the first 8 cycles and in combination with Rd from cycle 9 onwards.
  Interventions: Drug: Belantamab mafodotin; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone
- Cohort 8c: belantamab mafodotin 1.0 mg/kg Cycle 1,5;1.0 mg/kg Q9/12W from Cycle 9 +VRd/Rd (Experimental): Based on emerging data from Cohort 6-7, participants will receive 1.0 mg/kg IV dose of belantamab mafodotin on Day 1 of cycle 1 and cycle 5, then 1.0 mg/kg on day 1 of every third cycle from cycle 9 in combination with VRd for the first 8 cycles and in combination with Rd from cycle 9 onwards.
  Interventions: Drug: Belantamab mafodotin; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Belantamab mafodotin — Selected doses of belantamab mafodotin will be administered as intravenous infusion.
Drug: Bortezomib — Bortezomib will be administered subcutaneously or intravenously approximately 1 hour after the belantamab mafodotin infusion until Cycle 8.
Drug: Lenalidomide — Lenalidomide will be administered as 25 or 10 mg orally, depending upon renal function.
Drug: Dexamethasone — Dexamethasone will be administered orally as 20 mg in cycles 1-8 and 40 mg in Cycle 9 onwards.

SUMMARY:
This study will evaluate the safety, pharmacokinetics, pharmacodynamics and clinical activity of belantamab mafodotin in combination with Velcade (bortezomib), Revlimid (lenalidomide), dexamethasone (VRd) and will determine recommended phase 3 dose (RP3D) in adult participants with newly diagnosed multiple myeloma (NDMM). Participants will receive the combination of bortezomib, lenalidomide and dexamethasone (VRd) on a 3-week cycle until cycle 8, followed by the combination of lenalidomide and dexamethasone (Rd) on a 4-week cycle thereafter as per dosing schedule. Participants will receive belantamab mafodotin on a schedule that is dependent on the cohort to which they are assigned. Belantamab mafodotin will be administered in combination with VRd every 3 weeks (Q3W), every 6 weeks (Q6W), or every 9 weeks (Q9W) to Cycle 8, and then in combination with Rd every 4 weeks (Q4W), every 8 weeks (Q8W), or every 12 weeks (Q12W) thereafter. Participants will complete an End of Treatment (EOT) visit at the point of study treatment discontinuation, followed by a Safety Follow-up visit 70 days after EOT.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be over 18 years of age inclusive, at the time of signing the informed consent.
* Diagnosis of multiple myeloma with a requirement for treatment as documented per international myeloma working group (IMWG) criteria.
* Must have at least one aspect of measurable disease, defined as one of the following:
* Urine M-protein excretion >=200 mg/24 hours (>=0.2 gram [g]/24 hours), or
* Serum M-protein concentration >=0.5 grams per deciliter (g/dL) (>=5.0 gram per liter [g/L]), or
* Serum free light chain (FLC) assay: involved FLC level >=10 milligrams per deciliter (mg/dL) (>=100 milligram per liter [mg/L]) and an abnormal serum free light chain ratio (<0.26 or >1.65).
* Not a candidate for high-dose chemotherapy with autologous stem cell transplant (ASCT) due to presence of significant comorbid condition(s), such as cardiac, pulmonary or other major organ dysfunction that are likely to have a negative impact on tolerability of high dose chemotherapy with stem cell transplantation, as judged by the investigator.
* Eastern cooperative oncology group (ECOG) status of 0-2
* Adequate organ system functions as defined by the laboratory assessments listed as following: Absolute neutrophil count (ANC) >=1.5 x 10^9/L; Hemoglobin >=8.0 g/dL; Platelets >=75 x 10^9/L; Total bilirubin <=1.5 x upper limit of normal (ULN); (Isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%); Alanine aminotransferase (ALT) <=2.5 x ULN; eGFR >=30 mL/minute/1.73 meter^2; Urine Dipstick for protein OR Albumin/creatinine ratio (from spot urine)- Negative/trace (if >=1 plus only eligible if confirmed <=500 mg/gram (56 mg/millimoles [mmol]) by albumin/creatinine ratio (spot urine from first void); Left Ventricular Ejection Fraction (LVEF) by echocardiogram (ECHO) of >=35% participants with low LVEF (per institutional standards), consider referring to cardiology per local standards of care.
* Sex and Contraception/Barrier Requirements (Female):
* Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least 1 of the following conditions applies:
* Is NOT a woman of childbearing potential (WOCBP) or Due to lenalidomide being a thalidomide analogue with risk for embryofetal toxicity and prescribed under a pregnancy prevention/controlled distribution program, and bortezomib having the potential to cause fetal harm, WOCBP participants will be eligible if they commit to either: abstain continuously from heterosexual sexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR to use birth control as follows: Two methods of reliable birth control (one method that is highly effective and one additional effective (barrier) method), beginning 4 weeks prior to initiating treatment with lenalidomide, during therapy, during dose interruptions and continuing for 4 weeks following discontinuation of lenalidomide treatment. Thereafter, WOCBP participants must use one method of reliable birth control that is highly effective for a further 3 months following discontinuation of belantamab mafodotin, or a further 6 months following discontinuation of bortezomib, whichever is longer. WOCBP must also agree not to donate eggs (ova, oocytes) for the purpose of reproduction during treatment, during dose interruptions and for 28-days following the last dose of lenalidomide, 4 months following discontinuation of belantamab mafodotin treatment or 7-months following the last dose of bortezomib, whichever is longer. Two negative pregnancy tests must be obtained prior to initiating therapy. The first test should be performed within 10-14 days and the second test within 24 hours prior to prescribing the start of lenalidomide therapy.

The participant should not receive lenalidomide until the investigator has verified that the results of these pregnancy tests are negative. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention. The Investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.

* Sex and Contraception/Barrier Requirements (Male):
* Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
* Male participants are eligible to participate if they agree to the following from the time of first dose of study treatment until 28-days after the last dose of lenalidomide, 4-months after the last dose of bortezomib, or 6 months after the last dose of belantamab mafodotin, whichever is longer, to allow for clearance of any altered sperm: Refrain from donating sperm - Plus either: - Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR Must agree to use contraception/barrier as detailed below: Agree to use a male condom, even if they have undergone a successful vasectomy, and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year when having sexual intercourse with a WOCBP. Male participants should also use a condom when having sexual intercourse with pregnant females.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Smoldering multiple myeloma (SMM).
* Prior systemic therapy for multiple myeloma, or SMM. NOTE: An emergency course of steroids (defined as no greater than 40 mg of dexamethasone, or equivalent per day for a maximum of 4 days (that is, a total of 160 mg) is permitted. NOTE: Focal palliative radiation is permitted prior to enrollment, provided that it occurred at least 2 weeks prior to the first dose of study drug, that the participant has recovered from radiation-related toxicities, and that the participant did not require corticosteroids for radiation-induced adverse events.
* Participant is eligible for high dose chemotherapy with ASCT, as determined by a frailty score of 0 as assessed by the IMWG frailty index.
* Peripheral neuropathy or neuropathic pain Grade 2 or higher, as defined by the national cancer institute (NCI)-common terminology criteria for adverse events (CTCAE) Version 5.
* Major surgery within 4 weeks prior to the first dose of study drug.
* Presence of active renal condition (infection, requirement for dialysis or any other significant condition that could affect participant's safety). Participants with isolated proteinuria resulting from multiple myeloma (MM) are eligible, provided they fulfil criteria.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including lab abnormalities) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures.
* Evidence of active mucosal or internal bleeding uncontrolled by local therapy and not explained by reversible coagulopathy.
* Current active liver or biliary disease (except for Gilbert's syndrome or asymptomatic gallstones, or otherwise stable chronic liver disease as per the Investigator's assessment).
* Participants with previous or concurrent malignancies other than multiple myeloma are excluded. Exceptions are surgically treated cervical carcinoma in situ, or any other malignancy that has been considered medically stable for at least 2 years. The participant must not be receiving active therapy, other than hormonal therapy for this disease. Note: Participants with curatively treated non-melanoma skin cancer are allowed without a 2-year restriction.
* Evidence of cardiovascular risk including any of following: Evidence of current clinically significant untreated arrhythmias, including clinically significant electrocardiogram (ECG) abnormalities including second degree (Mobitz Type II) or third degree atrioventricular (AV) block; History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within 3 months of Screening.; Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system; Uncontrolled hypertension.
* Active infection requiring treatment.
* Known human immunodeficiency virus (HIV) infection.
* Presence of hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcAb), at Screening or within 3 months prior to first dose of study treatment.
* Positive hepatitis C antibody test result.
* Current corneal epithelial disease except for mild punctate keratopathy. Note: Participants with mild punctate keratopathy are allowed.
* Intolerance or contraindications to anti-viral prophylaxis.
* Unable to tolerate antithrombotic prophylaxis.
* AL amyloidosis (light chain amyloidosis), active polyneuropathy, organomegaly, endocrinopathy, monoclonal plasma proliferative disorder, skin changes (POEMS) syndrome or active plasma cell leukemia at the time of screening.
* Exhibiting clinical signs of or has a known history of meningeal or central nervous system involvement by multiple myeloma.
* Known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to drugs chemically related to belantamab mafodotin, or any of the components of the study treatment.
* Use of an investigational drug within 14 days or five half-lives (whichever is longer) preceding the first dose of study drug.
* Plasmapheresis within 7 days prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities (DLTs) | Treatment cycle 1 to 3 (each cycle of 21 days)
  The number of participants with DLTs will be reported.
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to an average of 54 months
  AEs and SAEs will be collected.

SECONDARY OUTCOMES:
Lenalidomide relative dose intensity (RDI ) of treatment with belantamab mafodotin in combination with VRd | 4 treatment cycles (each cycle of 21 days)
  RDI of treatment with belantamab mafodotin in combination with VRd will be analyzed.
Bortezomib RDI of treatment with belantamab mafodotin in combination with VRd | 4 treatment cycles (each cycle of 21 days)
  RDI of treatment with belantamab mafodotin in combination with VRd will be analyzed.
Cumulative administered dose of belantamab mafodotin treatment in combination with VRd | 4 treatment cycles (each cycle of 21 days)
  Cumulative administered dose of belantamab mafodotin in treatment in combination with VRd will be analyzed.
Maximum plasma concentration (Cmax) of belantamab mafodotin | Up to an average of 52 months
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Cmax of microtubule inhibitor monomethyl auristatin-F with a cysteine linker (cys-mcMMAF) | Up to an average of 52 months
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Area under the concentration time curve (AUC) of belantamab mafodotin | Up to an average of 52 months
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
AUC of cys-mcMMAF | Up to an average of 52 months
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Number of participants with positive anti-drug antibodies (ADAs) against belantamab mafodotin | Up to an average of 52 months
  Serum samples for the analysis of anti-belantamab mafodotin antibodies will be collected. The samples will be tested for anti-belantamab mafodotin antibodies using a tiered-testing scheme consisting of validated screening, confirmation, and titration assays.
Titers of ADAs against belantamab mafodotin | Up to an average of 52 months
  Serum samples for the analysis of anti-belantamab mafodotin antibodies will be collected. The samples will be tested for anti-belantamab mafodotin antibodies using a tiered-testing scheme consisting of validated screening, confirmation, and titration assays.
Overall Response Rate (ORR) | Up to 52 months
  ORR is defined as the percentage of participants with a confirmed partial response (PR) or better based on the response assessed by the investigator using International Myeloma Working Group (IMWG) criteria.
Complete Response Rate (CRR) | Up to 52 months
  CRR is defined as the percentage of participants with a confirmed complete response (CR) or better based on the response assessed by the investigator using IMWG criteria.
Rate of Very Good Partial Response (VGPR) or better | Up to 52 months
  Rate of VGPR or better is defined as the percentage of participants with a confirmed VGPR or better based on the response assessed by the investigator using IMWG criteria.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (28):
- United States (3):
  - GSK Investigational Site, Westwood, Kansas
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Madison, Wisconsin
- Australia (3):
  - GSK Investigational Site, Newcastle, New South Wales
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Fitzroy, Victoria
- Canada (2):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, London, Ontario
- GSK Investigational Site, Poitiers, France
- Germany (4):
  - GSK Investigational Site, Dresden
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Schwerin
  - GSK Investigational Site, Tübingen
- Italy (2):
  - GSK Investigational Site, Bologna
  - GSK Investigational Site, Meldola FC
- Poland (2):
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Poznan
- GSK Investigational Site, Seoul, South Korea
- Spain (7):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, PamplonaNavarra
  - GSK Investigational Site, Pozuelo de AlarcOn Madr
  - GSK Investigational Site, Santander
- United Kingdom (3):
  - GSK Investigational Site, Leicester
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com